CLINICAL TRIAL: NCT06749639
Title: An Open-Label, Single-Center, Dose-Escalation Clinical Study to Evaluate the Safety, Tolerability and Preliminary Efficacy of Intravitreal Injection of PUMCH-E101 in Subjects with RDH12 Retinopathy
Brief Title: Safety and Efficacy Study of PUMCH-E101 Injection in Subjects with RDH12 Retinopathy
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-E101
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Inherited Retinal Diseases
Keywords: Gene Therapy; Inherited Retinal Disease; RDH12 Mutations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PUMCH-E101 Treatment Arm（Low dose） (Experimental): Intraocular injection of a single low dose of PUMCH-E101
  Interventions: Genetic: PUMCH-E101 Injection（Low dose）
- PUMCH-E101 Treatment Arm（High dose） (Experimental): Intraocular injection of a single high dose of PUMCH-E101
  Interventions: Genetic: PUMCH-E101 Injection（High dose）

INTERVENTIONS:
Genetic: PUMCH-E101 Injection（Low dose） — Single intravitreal injection
  Arms: PUMCH-E101 Treatment Arm（Low dose）
Genetic: PUMCH-E101 Injection（High dose） — Single intravitreal injection
  Arms: PUMCH-E101 Treatment Arm（High dose）

SUMMARY:
The goal of this clinical trial is to evaluate the safety and efficacy of PUMCH-E101 injection in subjects with RDH12 retinopathy.

DETAILED DESCRIPTION:
This is an open-label, single-center, dose-escalation study. One eye of each participant will receive a single intravitreal injection of PUMCH-E101. Participants will be followed for 52 weeks after which they will continue to be followed for up to 5 years after enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily participate and sign the informed consent form;
2. Age between 8-45 years old, gender is not limited;
3. Clinical diagnosis of IRD caused by RDH12 mutations;
4. The Best Corrected Visual Acuity (BCVA) detected by the Early Treatment Diabetic Retinopathy Study (ETDRS) eye chart in the study eye is less than or equal to 63 letters, which is equivalent to 20/63 of the Snellen Eye Chart;
5. At screening, the blood pregnancy test result of females of childbearing potential (e.g., females who have not undergone surgical sterilization or less than 1 year after menopause) is negative. Male and female subjects of childbearing potential agree to use effective contraception throughout the study and for at least 12 months after dosing.

Exclusion Criteria:

1. Opacity of refractive media or inability to dilate pupils in the study eye that significantly interferes with visual acuity detection, anterior segment or fundus assessment;
2. Presence of diabetic retinopathy, retinal vein occlusion, pathological myopia, retinal detachment, or other conditions in the study eye that are assessed by the investigator as affecting the safety of the subject or the validity of the study;
3. Any intraocular surgery in the study eye within 3 months prior to screening;
4. Active intraocular or periocular infection (such as blepharitis, conjunctivitis, keratitis, scleritis, etc.) in the study eye;
5. History of uveitis in either eye；
6. Those with diffuse intravascular coagulation and obvious bleeding tendency (such as hemoptysis, hematemesis, severe purpura, etc.) within 3 months before screening;
7. History of myocardial infarction, unstable angina, coronary revascularization, cerebrovascular accident (including TIA), history of other thromboembolic diseases (such as thromboembolic angiitis, pulmonary embolism, deep vein thrombosis, portal vein thrombosis, etc.), New York Heart Association (NYHA) grade ≥ II cardiac insufficiency, severe unstable ventricular arrhythmia, within 6 months prior to screening;
8. Subjects with systemic immune diseases (including systemic lupus erythematosus, ankylosing spondylitis, rheumatoid arthritis, etc.);
9. Diabetic patients with any of the following conditions: Known macrovascular complications or Glycosylated hemoglobin at screening（HbA1c）>7.5% or Those who have received more than two oral hypoglycemic drugs or received insulin or GLP-1 receptor agonists therapies;
10. Hypertensive patients with poor blood pressure control (defined as: systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥100 mmHg when the subject is seated after receiving antihypertensive medication);
11. Any uncontrollable clinical illness (such as severe psychiatric, respiratory and other systemic diseases and history of malignant tumors);
12. Subjects with abnormal liver and kidney function: alanine aminotransferase (ALT)/aspartate aminotransferase (AST) ≥ 2 times the upper limit of normal; Total bilirubin ≥ 1.5 times the upper limit of normal, creatinine and urea/urea nitrogen ≥ 1.5 times the upper limit of normal;
13. Subjects with abnormal coagulation function: prothrombin time (PT) > upper limit of normal value of 3 seconds or activated partial thromboplasting time (APTT) > upper limit of normal value of 10 seconds; Haemoglobin (HGb) < 10 g/dL;
14. Those who are positive for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, treponema pallidum antibody and human immunodeficiency virus (HIV) antibody;
15. Those who are known to be allergic to the therapeutic drugs or diagnostic drugs used in the study protocol, including the investigational products, etc.;
16. Those who have used anticoagulant or antiplatelet drugs within 7 days before dosing;
17. Currently using or may need to use drugs that can cause crystalline toxicity or retinal toxicity (such as deferoxamine, chloroquine/hydroxychloroquine, tamoxifen, ethambutol, etc.);
18. Those who have a history of surgical operation within 1 month before screening, and/or currently have unhealed wounds (wound degree> stage III), moderate to severe ulcers, and fractures;
19. Subjects with systemic infectious diseases requiring systemic treatment (oral, intramuscular or intravenous) at the time of screening;
20. Those who have received any AAV gene therapy products in the past;
21. Pregnant or lactating females;
22. Those who have participated in any clinical trial of drugs (excluding vitamins and minerals) within 3 months before screening;
23. Other individuals who need to be excluded, as determined by the investigator

Ages: 8 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-09-20 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2030-01-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of DLTs | 4 weeks
  Number and proportion of dose limited toxicity (DLTs)
Incidence of AEs | 52 weeks
  Number and severity of overall and ocular Adverse Events (AEs)
Incidence of SAEs | 52 weeks
  Number and severity of overall and ocular Serious Adverse Events (SAEs)

SECONDARY OUTCOMES:
Visual function | 52 weeks
  Change from baseline in BCVA (Best Corrected Visual Acuity) (ETDRS)
Visual function | 52 weeks
  Change from baseline in the mean value of the photosensitivity threshold (Full-field Threshold)
Visual function | 52 weeks
  Change from baseline in mean sensitivity (MS) (Static visual field)

CONTACTS AND LOCATIONS:
Overall Officials: Ruifang Sui, MD, PhD, Principal Investigator — Peking Union Medical College Hospital, Department of Ophthalmology
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No